CLINICAL TRIAL: NCT06440148
Title: Role of Sclerostin in Mastocytosis Bone Disease
Brief Title: Relationship Between Circulating Sclerostin and Bone Lesions in Patients With Mastocytosis
Status: Recruiting | Type: Observational
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Aneta Szudy Szczyrek, Doctor of Medicine, Medical University of Lublin
Other Study IDs: SCLERMAST01
Record Dates: First submitted 2024-05-06; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Mastocytosis; Bones
Keywords: Bones; Mastocytosis; Osteolysis; Osteosclerosis; Sclerostin
MeSH Terms: conditions — Mastocytosis; Osteolysis; Osteosclerosis; Sclerosteosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The studied material is approximately 2.5 ml of peripheral blood collected into plasma gel tubes.
  The samples are centrifuged at 3000 rpm for 10 min, plasma is pipetted into tubes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: SCLEROSTIN — Pathogenesis of mastocytosis bone disease

SUMMARY:
Mastocytosis is very rare and highly heterogeneous group of disorders, characterized by the accumulation of clonal mast cells which can infiltrate several organs and tissues.

Bones are the most frequent localization of systemic mastocytosis. The aim of our research was to explain the potential role of sclerostin in the pathogenesis of bone disease in mastocytosis.

DETAILED DESCRIPTION:
Mastocytosis is a heterogeneous group of disorders, characterized by the accumulation of clonal mast cells which can infiltrate several organs, such as the skin, bone marrow or liver. The skeleton is the most frequent localization of systemic mastocytosis (SM). Bone involvement occurs in approximately 70% of SM patients. Pathogenesis of mastocytosis bone disease is poorly understood.

The aim of our research is to explain the potential role of sclerostin, a recently discovered bone tissue protein, in the pathogenesis of bone changes in patients with mastocytosis.

The study group consists of adult patients with mastocytosis divided according to their clinical variants of disease (aggressive systemic mastocytosis - ASM, systemic mastocytosis with an associated hematological neoplasms SM-AHN, smouldering systemic mastocytosis - SSM, indolent systemic mastocytosis - ISM and cutaneous mastocytosis - CM; and group of healthy volunteers.

The concentration of sclerostin, bioactive sclerostin and expression of the SOST gene in human plasma and HMC-1.2 human mast cell culture supernatants is assessed. The Real-Time PCR method is used to evaluate the expression of sclerostin at the mRNA level, while the concentration of the sclerostin protein and its bioactive form is assessed using the enzyme immunoassay ELISA method. The obtained results are correlated with selected demographic, clinical, laboratory and radiological findings. Low-dose CT scan is used to assess bone changes.

These preliminary results could serve that sclerostin may be a new therapeutic target in patients with mastocytosis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Mastocytosis defined according to WHO criteria
* Known KIT mutation status

Exclusion Criteria:

* History of organ transplant
* Inability to give informed consent
* Pregnancy, Breastfeeding
* Vulnerable Patient, defined as: patient with another uncontrolled severe disease; patient under juridical protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study group consists of adult patients diagnosed with mastocytosis, divides according to the clinical variants: aggressive systemic mastocytosis (ASM), systemic mastocytosis with associated hematological neoplasm (SM-AHN), indolent systemic mastocytosis (ISM), smoldering systemic mastocytosis (SSM) and cutaneous mastocytosis (CM).
  The diagnosis of mastocytosis should be established based on biopsy of the affected organ (bone marrow trephine biopsy, skin affected by the disease), following the 2022 WHO classification. The control group comprised 30 healthy volunteers matched with the study group in terms of age and gender.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
plasma sclerostin measurements (in pmol/l) SOST gene expression by Real-Time PCR dimensions of osteolytic lesions on low-dose computed tomography (in mm) dimensions of osteosclerotic lesions on low-dose computed tomography (in mm) | 1 year
  The Primary Outcome Measures concern:
  * the measurements of plasma levels of sclerostin and its bioactive form in patients with mastocytosis and healthy volunteers
  * the measurements of levels of sclerostin and its bioactive form in HMC-1.2 human mast cells unstimulated and stimutaled with Il-6
dimensions of osteolytic lesions (in mm) | 1 year
  The Primary Outcome Measures concern:
  - the measurements of the dimensions of osteolytic bone lesions on low-dose computed tomography in patients with mastocytosis
dimensions of osteosclerotic lesions (in mm) | 1 year
  The Primary Outcome Measures concern:
  - the measurements of the dimensions of osteosclerotic bone lesions on low-dose computed tomography in patients with mastocytosis

CONTACTS AND LOCATIONS:
Overall Officials: Aneta A Szudy-Szczyrek, MD., PhD., Principal Investigator — Medical University of Lublin
Locations (1):
- Department of Hematooncology and Bone Marrow Transplantation, Lublin, Lublin Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided